CLINICAL TRIAL: NCT06689904
Title: The Effect of Eyedrop Size on Pupillary Dilation Using the Nanodropper Bottle Adapter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sutter Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1826733-1
Record Dates: First submitted 2024-11-07; First posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Medication Delivery; Eye Drop Delivery
Keywords: eye drops; pupil dilation; eye drop bottle device; eye drop size
MeSH Terms: conditions — Mydriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Eye dilated with the nanodropper (Experimental): For each participant, one eye (left or right) is randomly selected to be dilated with the Nanodropper.
  Interventions: Device: Nanodropper
- Eye dilated with the standard bottle (Active Comparator): Fellow eye is dilated with the standard eye drop bottle
  Interventions: Device: Standard eye drop bottle

INTERVENTIONS:
Device: Nanodropper — One eye is randomly selected to be dilated with the nanodropper
  Arms: Eye dilated with the nanodropper
Device: Standard eye drop bottle — eye is dilated with the standard eye drop bottle
  Arms: Eye dilated with the standard bottle

SUMMARY:
The average drop size produced by standard eyedrop bottle exceeds the maximal capacity that the human eye are absorb topically. This excess leads to medication waste, increased costs, and greater risk of side effects.

The Nanodropper is a commercially available, FDA listed eyedrop bottle adapter that delivers a smaller drop size. The investigators hypothesize the Nanodropper is noninferior to the standard eye drop bottle for pupil dilation.

In this study, participants have one eye randomly chosen to be dilated with the Nanodropper and the fellow eye dilated with the standard bottle with a 50/50 mixture of tropicamide 1% and phenylephrine 2.5%. Pupil size before and after 30 minutes of dilation are measured with a pupillometer and compared between fellow eyes to see if there is a difference.

DETAILED DESCRIPTION:
Ophthalmic medications are available in eyedrop bottles that produce on average a drop size of about 40 uL, while the human eye can only hold about 7-10uL. This excess leads to medication waste, increased costs, and greater risk of side effects.

The Nanodropper is a commercially available, FDA listed (class 1 medical device, 510(k) exempt) eyedrop bottle adapter that delivers a smaller drop size of 10 uL. The investigators hypothesize the Nanodropper is noninferior to the standard eye drop bottle for pupil dilation.

This is a prospective comparative matched pairs study of adults scheduled for routine bilateral eye dilation. Exclusion criteria includes anisocoria and medications affecting pupil size. One eye is randomly dilated with the Nanodropper and the fellow eye dilated with the standard bottle with a 50/50 mixture of tropicamide 1% and phenylephrine 2.5%. Pupil size before and after 30 minutes of dilation are measured with a pupillometer and compared between fellow eyes within the same subject with a noninferiority margin of 0.5mm.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years old
* scheduled for routine bilateral eye dilation

Exclusion Criteria:

* narrow angles
* allergies to phenylephrine or tropicamide
* concurrent use of any mydriatic agents (e.g., atropine, cyclopentolate, brimonidine)
* baseline anisocoria (>1 mm)
* traumatic pupil,
* surgical pupil
* unilateral pseudoexfoliation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2022-01-04 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Pupil size (diameter) | 30 minutes after dilation
  Pupil diameter (mm)

CONTACTS AND LOCATIONS:
Locations (1):
- Lions Eye Clinic, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No